CLINICAL TRIAL: NCT06894940
Title: Rehabilitation of the Upper Limb in Progressive Multiple Sclerosis: a Clinical and MRI Study of Different Rehabilitative Protocols in Patients Treated with Anti B Monoclonal Antibodies
Brief Title: Rehabilitative Protocols in Progressive Multiple Sclerosis Treated with Anti CD20 Monoclonal Antibodies
Acronym: Reup
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pavia (Other)
Collaborators: University of Genova (Other); Consorzio per Valutazioni Biologiche e Farmacologiche (Other); A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Antonio Nardone, prof, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF-2019-12370447
Record Dates: First submitted 2025-03-12; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Task oriented rehabilitation with virtual reality (Experimental): The intensive task oriented physiotherapy consists of focused single tasks (reaching a glass on the table) and occupational therapy on activities (tasks). The VR BTS NIRVANA system allows the patient to interact with virtual reality scenarios associated with daily activity tasks with increasing levels of complexity. NIRVANA is a system that projects on the wall or on the floor a large scenario where an interactive series of exercises is reproduced.In this project, the categories of exercise are 1.Sprites: patient is required to reach, touching or grabbing a series of objects. 2.Follow me: patient is required to control movement. 3.Motion: patient is required to focus on the quality of movement. 4.Hunt: patient is required to reach objects 5.Games: includes a list of effects that can be used by the therapist to define new personalized exercises.
  Interventions: Behavioral: Experimental
- Task oriented rehabilitation (Active Comparator): ntensive task oriented physiotherapy and occupational therapy of the upper limb, once every day, 3 hours a day for 4 weeks.
  Interventions: Behavioral: Active Comparator #1
- Passive mobilization (Placebo Comparator): The passive mobilization protocol consists of passive movements of the proximal and distal parts of the upper limbs
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Active Comparator #1 — task oriented rehabilitation
  Other Names: task oriented rehabilitation
  Arms: Task oriented rehabilitation
Behavioral: Placebo — passive rehabilitation
  Other Names: passive rehabilitation
  Arms: Passive mobilization
Behavioral: Experimental — rehabilitation with virtual reality
  Other Names: rehabilitation with virtual reality
  Arms: Task oriented rehabilitation with virtual reality

SUMMARY:
Progressive multiple sclerosis (MS) patients have usually a worsening clinical course and it remains unclear if rehabilitation can indeed slow down the progression of the disease. Recently, clinical studies demonstrated that a treatment with monoclonal antibodies against B lymphocytes can have a positive effect on the progression of disability. Therefore now the investigators have, in this phase of the disease, a treatment that can impact the clinical course, even if the effect is not complete. The present study project has the aim to verify if, in progressive MS treated with monoclonal antibodies, a high technology rehabilitative protocol added to an intensive rehabilitation program is more effective on the motor recovery, in particular of the upper limb, as compared to an intensive traditional scheme of rehabilitation and to a passive treatment therapy, Moreover, the MRI functional reorganization of the central nervous system will be evaluated as well as the duration of the rehabilitative effect.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune inflammatory disease of the central nervous system that cause relevant disability, but also personal and familial suffering. Usually, after 10-15 years from the onset, the disease acquires a progressive clinical course or alternatively the progressive onset can open the disease, in 10-15% of cases. When MS has entered the progressive course, the disorder can be clinically active with relapses or progression, or with MRI signs of activity such as the presence of Gadolinium enhancing lesions, new T2 or enlarging lesions. While in the relapsing remitting phase (RR) of the disease inflammation is the main neuropathological process, in the progressive phase of the disease other mechanisms certainly occur, such as degeneration of the previously damaged neurons and axons. In the RR course of MS the investigators have numerous different treatments that are, in the majority of cases, efficacious. On the contrary, when the disease assumes a progressive course, the treatments are usually ineffective and also the effectiveness of rehabilitative treatments are of uncertain utility. Moreover, this population of patients is usually characterized at MRI by a relevant lesion load that could have a negative effect on the plasticity properties of a heavily damaged central nervous system. Recently, clinical studies demonstrated that a treatment with monoclonal antibodies against B lymphocytes can have a positive effect on the progression of disability. The results of this study indicate that now the investigators have, in this phase of the disease, a treatment that can impact the clinical course, even if the effect is not complete. In the progressive MS the main problem is usually the loss of strength in the lothe investigatorsr limbs, with difficulty in walking and balance. The pyramidal tracts are lesioned at different numerous levels and the axons with a longer length show widespread processes of Wallerian degeneration, that at the moment the investigators cannot reverse. Also the upper limbs are hothe investigatorsver affected, but have a higher probability to be less injured and damaged, with a resulting possibility to partially recover with an appropriate rehabilitative treatment. There are studies that report a high percentage of upper limb dysfunction, not only in progressive phase of the disease but also in early stage of the disorder. The efficacy of medical therapy and/or rehabilitation in upper limb dysfunction in MS is not clear. This question is relevant for the importance of upper limb function in order to retain an acceptable level of independence. In these last years a systematic review on upper limb rehabilitation in multiple sclerosis was published. This review provides an analysis of the upper limb rehabilitation strategies in persons with MS, evaluating thirty articles that met the criteria for data extraction. The conclusions of the review are that different types of rehabilitation strategies can improve upper limb function, but further research is necessary to compare directly the effects of different rehabilitation strategies and to investigate the optimal therapy dosage according to the upper limb disability level. The investigators recently investigated the problem of upper limb rehabilitation in progressive MS, demonstrating that an active rehabilitation treatment improves several motor tasks and increased the cerebral connectivity, especially in the cerebellar and thalamic networks. In the present research project the investigators have the aim to study if an innovative medical therapy associated to an intensive high technology rehabilitative protocol has the capacity to ameliorate further the upper limb function and to influence the central nervous system reorganizing networks.Hyphotesis and Significance: It is possible that in progressive MS cases, treated with anti B monoclonal antibodies, and therefore in cases where the inflammatory component of the disease is partially under control, a rehabilitative therapy could be more effective than in cases that are not treated and where the disorder has a not modifiable worsening clinical course. The investigators will evaluate in this particular population of patients if a high technology protocol with virtual reality added to an intensive traditional rehabilitative treatment can induce an improvement of the motility in the upper limb as compared to the traditional intensive therapy and to a passive mobilization regimen. Also the functional MRI reorganization could be different in the treated groups. The final target of the project is to demonstrate that also in the progressive phase of the disease a medical therapy associated to an innovative rehabilitation protocol has the capacity to improve the motor activity in the upper limb and that this treatment has an impact also on the functional reorganization of the central nervous system, at least for a period of time.

Preliminary Data:

Recently the investigators evaluated a small population of MS patients with a progressive clinical course of disease (26 cases not receiving any disease modifying therapy) and treated with an active occupational rehabilitative protocol as compared to a passive mobilization therapy. All the cases have also been examined with functional and structural MRI. The results show that both treatments have the capacity to improve the upper limb motor activity, and the difference between the two diverse protocols the investigators are not significant in a few motor tasks. The improvement of the 9 Hole Peg test (9HPT) in the active treatment was of 2.1 seconds as compared to baseline, that was almost significant (p= 0,06) if compared to the passive treatment group. On the contrary, if the distal upper limb motility was evaluated with an engineered glove a difference between the two different treatment protocols was detected. Moreover, the active occupational therapy had the capacity to induce relevant modification in the functional cerebral networks detected at MRI, with an increase of connectivity between cerebellar and thalamic networks in the actively treated patients (5).Specific Aim 1: The aim 1 of the present research project is to characterize and compare, in progressive MS cases patients treated with monoclonal anti B antibodies, the effect of different rehabilitative protocols on the motor activity in the upper limb trough clinical and functional evaluations .The patients will be randomized in a passive treatment group, in an intensive standard rehabilitative protocol or in an intensive standard rehabilitative protocol plus a high technology treatment with virtual reality.

The influence of these different rehabilitative treatments on manual dexterity and upper limb function will be examined and compared. Patients will be evaluated at baseline, at the end of the treatment and after 3 months with scales and tests specifically addressed to examine the upper limb motility. Moreover the investigators will utilize also an engineered glove that has the capacity to detect light motor impairment in the finger movements, especially in the bimanual coordination setting.The aim 2 is to improve the general neurological condition of the patient. All the MS cases, beyond the rehabilitative protocols mainly focused on the upper limb, will receive also a complete rehabilitation program, addressed on balance, gait, posture, fatigue and cognition. The aim 3 is to evaluate if a rehabilitative program can also induce a partial reorganization of the central nervous system.

Resting state, functional MRI and diffusion tensor imaging are utilized in order to detect the changes that different rehabilitative protocols can determine on brain functioning, brain connectivity and structural integrity of the white matter tracts. There are few studies that addressed the effect of rehabilitation on MRI, demonstrating an improved integrity of the corpus callosum or changes in the microarchitecture of white matter tracts , or functional and structural modification after motor rehabilitation programs. However the majority of these studies have been carried out in the RR phase of the disease and is unclear if in progressive forms of MS the damaged central nervous system has the capacity to improve its functional connectivity or to partially repair the nervous system structure.

ELIGIBILITY:
Inclusion criteria:

* age 25-65 years;
* right-handed
* progressive active form of MS treated with anti B monoclonal antibodies, Ocrelizumab or Rituximab since at least 6 months.
* EDSS 3-7.
* absence of relevant cognitive deficiency, as evaluated with Brief International Cognitive Assessment for MS (Bicams) °absence of visual or audio deficit disorders.

Exclusion criteria:

* history of a cardiovascular disorder or any other disease that can hamper the active participation to the research project.
* Contraindication to perform MRI exams

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
The Primary endpoint is the improvement in the distal motility of the upper limb evaluated with the Nine Hole Peg test. | baseline and after 2 and 5 months
  It explores distal upper limb motility and is evaluated in seconds, with higher values corresponding to worse perfomance

SECONDARY OUTCOMES:
Patients will be evaluated at baseline, at the end of the treatment period and after 3 months with the the action research arm test (ARAT). | at baseline, after 2 and 5 months
  Specific test for proximal and distal upper limb motility. It ranges from 0 to 57 and higher values indicating better performance

CONTACTS AND LOCATIONS:
Overall Officials: antonio nardone, prof, Principal Investigator — University of Pavia
Locations (1):
- ICS Salvatore Maugeri, Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No